CLINICAL TRIAL: NCT02536872
Title: An Observational Study of the Effect of Antibiotics on the Microbiology of the Bladder in Patients With Overactive Bladder
Brief Title: A Study of the Effect of Antibiotics on the Microbiology of the Bladder in Patients With Overactive Bladder
Status: Completed | Type: Observational
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Jonathan Duckett, Consultant Urogynaecologist, Medway NHS Foundation Trust
Other Study IDs: 19/06/2015
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Urogynaecology
Keywords: infection overactive bladder
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: None - this is a prospective observational study. Patients will be prescribed their usual treatment (antibiotics) and the effect on urine studied

SUMMARY:
The concept of organisms living on or in the human body without causing overt signs of an infection is common in medicine and has been termed a microbiome. Urine from patients with Overactive bladder (OAB) grows different organisms from controls without OAB. However, it is not known if the bacteria that have been identified are innocent commensals or pathogenic organism responsible for the symptoms of OAB. Previous data suggests that treatment with antibiotics does lead to an improvement in overactive bladder symptoms in a large number of patients. On this basis the investigators now treat are patients with similar antibiotic regimes. If antibiotics improve symptoms it would be expected that they would return the microbiome back to how it is in patients without OAB. This study aims to identify the effects of antibiotics on the urinary microbiome and to identify/confirm if antibiotic treatments cause improvement in OAB.

DETAILED DESCRIPTION:
This study is a consecutive cohort study. Subjects will be recruited from Urogynaecology clinics at Medway NHS Foundation Trust. Patients will be identified from previous records and also prospectively from new patients. They will be sent information regarding the trial before attending their first appointment.

Patients attending urogynaecology clinics will provide a fresh clean catch specimen of urine. A conventional hospital Mid stream speciemn of urine (MSU) will be sent. Urine will be dipsticked for nitrites and leucocyte esterase. The urine will then be spun and undergo microscopy using a special stain (looking for intracellular organisms in shed urothelial cells). The urothelial cells will be cleaned with antibiotics. The cells will then be lysed and their contents cultured. The contents will undergo Polymerase Chain Reaction (PCR) sequencing to identify bacteria. Sensitivity testing will be used to assess and deliver the appropriate antibiotic regime.

Women will be treated with a 6 week course of antibiotics as per their usual treatment. Broad spectrum antibiotics will be prescribed to all women based on the previous successful therapeutic regime as described by Vijaya. Six weeks after the end of antibiotic therapy patients will be reviewed and their urine retested.

ELIGIBILITY:
Inclusion Criteria:

1. > age 18 years
2. Negative urine dipstick (nitrites) and culture (x10 to the power 5 colony forming units) x105 cfu
3. Idiopathic overactive bladder as per International Continence Society definition

Exclusion Criteria:

1. Patients treated with antibiotics for any infection within the last 6 weeks.
2. Patients with known multiple sclerosis, stroke, spinal injury, or other neurological disease
3. Urinary tract infection diagnosed by nitrite positivity or positive urine culture (x105 cfu)
4. Undiagnosed macroscopic or persistent microscopic haematuria needing investigation
5. Previous or current cancer of the urogenital tract.
6. Contraindication to multiple antibiotics
7. No suitable oral antibiotic regime
8. Patients unable to understand the study or complete the questionnaires.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with overactive bladder syndrome
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in bladder microbiology in patients treated with antibiotics. | 6 weeks
  The number and type of different organisms will be quantified and compared to the pre treatment organisms

SECONDARY OUTCOMES:
Change in the overactive bladder questionnaire (OAB-q) before and after treatment | 6 weeks
  questionnaire
Change in Patient Perception of Bladder Condition (PPBC) | 6 weeks
  questionnaire
To identify adherence to the treatment regime | 6 weeks
  Patients will be asked to identify if they took all of the antibiotics; 75% of the time; 50 or 25%
To identify adverse effects of the treatment | 6 weeks
  Patients will be asked report side effects of antibiotic treatment
Changes in symptoms using (change from baseline to assessment) | 6 weeks
  Measured by the International consultation on Incontinence female lower urinary tract syptome questionnaire. (ICI FLUTs)

CONTACTS AND LOCATIONS:
Locations (1):
- Medway Hospital, Gillingham, Kent, United Kingdom